CLINICAL TRIAL: NCT05351489
Title: Effect of Two Different Doses of Intrathecal Dexmedetomidine as Adjuvant Combined With Hyperbaric Bupivacaine in Elderly Patients Undergoing Transurethral Resection of Prostate: A Prospective, Randomized Study
Brief Title: Effect of Two Different Doses of Intrathecal Dexmedetomidine as Adjuvant in Elderly Patients Undergoing HoLEP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mahmoud Mahmoud Othman, Clinical professor of anesthesia and surgical Intensive care, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MS.22.04.157
Record Dates: First submitted 2022-04-17; First posted 2022-04-28 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Transurethral Resection of Prostate
MeSH Terms: interventions — Dexmedetomidine; Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: double- blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine 5 μg group (D5 group ) (Experimental): Dexmedetomidine 5 μg group (D5 group ): Patients will receive 2 mL heavy bupivacaine 0.5% and Dexmedetomidine 5 μg intrathecal.
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine 10 μg group (D10 group ) (Active Comparator): dexmedetomidine 10 μg group (D10 group ): Patients will receive 2 mL heavy bupivacaine 0.5% and Dexmedetomidine 10 μg intrathecal .
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Patients will receive intrathecal 2 mL heavy bupivacaine 0. 5% together with either dexmedetomidine 5 μg or10 μg dexmedetomidine .
  Other Names: Group (D 5):Patients will receive intrathecal 2 mL heavy bupivacaine 0. 5% together with dexmedetomidine 5 μg dexmedetomidine .; Group (D10):Patients will receive intrathecal 2 mL heavy bupivacaine 0. 5% together with dexmedetomidine 10 μg dexmedetomidine

SUMMARY:
Transurethral resection of the prostate (TURP) is the most common Surgical intervention for elderly patients with benign prostatic hyperplasia. Spinal anesthesia is the technique of choice in TURP.Intrathecal (IT)adjuvants prolong the duration of spinal anesthesia and postoperative analgesia there by reducing the requirement of postoperative supplement analgesics .The incorporation of adjuvants also lowers the overall dose of local anesthetic and associated side effects .

The extended analgesic efficacy of intratheacal dexmedetomidine in the postoperative period has been shown in a few clinical studies . These authors have studied different doses (2 - 10 μg) of intrathecal dexametomedine and compared it with various other adjuvants like clonidine, fentanyl, midazolam, buprenorphine, etc., with varying results . The existing studies comparing different doses of intratheacal dexmedetomidine are few. Moreover none of these studies have stressed the dose-response relationship between different doses of intratheacal dexmedetomidine and differential analgesia (DA) defined as the time difference from the offset of motor blockade to the first analgesic requirement on numerical rating scale more than4.

DETAILED DESCRIPTION:
The study hypothesis is that there may be a dose dependent prolongation of dexametomedine with escalating doses of intrathecal dexmedetomidine.In this study we tried to find out the optimum safe dose of dexametomedine that used as adjuvant with bupivacaine for patient undergoing transuretheral reseaction of large sized prostate.

The aim of the current study is to To elucidate the dose-response relationship between intrathecal dexametomedine with different doses and subarachnoid block characteristics, particularly the duration of analgesia and differential analgesia. Considering the dose dependent action of intrathecal dexametomedine, the authors could hypotheize that the higher dose of dexametomedine (10 μg) used as adjuvant with bupivacaine will result in better efficacy profile with further prolongation of sensory motor blockade in elderly patient undergoing transurethral resecation of large sized prostate if compared with dexametomedine (5 μg).

After obtaining approval from Mansoura Faculty of Medicine Institutional Research Board about This study which will be a double blinded, prospective, randomized, trial. This study will be carried out in the Urology and Nephrology center of Mansoura university (MUCH). An informed written consent will be obtained from all patient.

This study will be conducted on 70 patients 55- 85 years of age, American Society of Anesthesiologists (ASA) physical status I/II scheduled for transurethral reasection of prostate .

The study subjects will be randomly assigned to one of two equal groups (dexmedetomidine5 μg group and dexmedetomidine 10 μg group ) using computer generrated randomization members Dexmedetomidine 5 μg group (D5 group ): Patients will receive 2 mL heavy bupivacaine 0. 5% and Dexmedetomidine 5 μg dexmedetomidine 10 μg group (D10 group ): Patients will receive 2 mL heavy bupivacaine 0. 5% and Dexmedetomidine 10 μg All patients will be subjected to preoperative assessment that includes thorough clinical examination, radiological and laboratory workup. Laboratory investigations will include complete blood count (CBC), serum electrolytes, arterial blood gas, urine analysis, coagulation survey, blood glucose level, liver and renal function tests. ECG, transthoracic echocardiography and chest x-ray will be done.

All patient will be hospitalized at least a day before surgery and will be kept nil per os for 8 hours.Before the procedure the investigator will measure and record baseline heart rate (HR) and mean arterial pressure (MAP) will be assessed by noninvasive blood pressure monitoring, as well as arterial oxygen saturation, then all participants will be received 10 mL/kg of crystalloid (Ringer's solution) in the supine position on arrival to the operating room, and finally divided into two groups using block randomization: SA will be performed with a 22-25-gauge Quincke needle at the L3/L4 or L4/L5intervertebral space The first group (dexmedetomidine5 μg group) will be received 2mL (10 mg) of heavy bupivacaine plus 5 μg of dexmedetomidine intrathecally in 1 ml insulin syringe the second (dexmedetomidine 10 μg group),will be received 2 mL (10 mg) of heavy bupivacaine plus 10 μg dexmedetomidine in 1 ml insulin syringe.

The duration of analegesia will be investigated.Also,Total dose of analgesic requirements 24 hrs postoperative),Intra operative heart rate and blood pressure every 15 min till the end of surgery,Postoperative blood pressure and heat rate at 2,4,6,12 and 24 hour ,Onset of sensory block after spinal anesthesia (minute),Onset of motor block after spinal anesthesia (minute),Time to achieve sensory block at T8 or higher dermatome (using pin prick test every 1 minute) (minute),Time to achieve sensory block level at T12 and L1 dermatomes and spinal anesthesia wearing off (minute),Dose of vasopressors required

,Visual analog scale Immediately Recovery and 2,4,6 and 12 hours after operation Differenrtial analgesia (time difference from the offset of motor blockade to the first analgesic required ).Postoperative complications (nausea, vomiting, pruritis, hypotension and shivering )will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Elderly patients undergoing transurtheral resection of Prostate.
2. American Society of Anesthesiologists (ASA) physical status I/II

Exclusion Criteria:

1. Any contraindication to subarachnoid block.
2. On chronic analgesic therapy.
3. Patients refuse to contribute in the study.
4. Cognitive impairment.
5. Not able to understand numerical rating pain scale (NRS). 6.-Significant comorbid conditions like uncontrolled hypertension, congestive heart failure myocardial infarction in the past 6 months..

Ages: 60 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Study will carried out for elderly male patients undergoing transuretheral resection of prostate.
Enrollment: 70 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The duration of analgesia | perioperative time for 24 hours
  Duration of spinal analgesia till analgesic rescue.

SECONDARY OUTCOMES:
Total dose of analgesic requirements . | perioperative time for 24 hours
  Record the total analgesic rescue to allow visual analogue score less than3
Hemodynamic stability perioperatively. | perioperative time for 24 hours
  Intra operative systolic and diastolic arterial blood pressure every 15 min till the end of surgery.Postoperative systolic and diastolic arterial blood pressure at 2,4,6,12 and 24 hour
Onset of sensory block after spinal anesthesia . | Immediate after spinal anesthesia
  Onset of sensory loss after spinal anesthesia in minutes.
Dose of vasopressors required | perioperative time for two hours postoperatively
  Dose of ephedrine or norepinephrine used to counteract any hypotension.
Perioperative hypotension | Perioperative time for 24 hours postoperatively
  Record number of patients with any drop of systolic blood pressure below 90 mmHg
Differential analgesia | Perioperative time for 24 hours.
  Record the time difference from the offset of motor blockade to the first analgesic required

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud M Othman, MD, Principal Investigator — Department of anesthesia ,Urology and nephrology center ,Faculty of medicine,Mansoura university; Taha R Elashmawy, BCH, Study Chair — Department of anesthesia ,Urology and nephrology center ,Faculty of medicine,Mansoura university
Locations (1):
- Urology and nephrology center, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: One year
Access Criteria: Pubmed